CLINICAL TRIAL: NCT04479215
Title: Postoperative Feeding Practice and Its Effect on Postoperative Vomiting in Children Undergoing Infra-umbilical Daycare Surgery: A Prospective Observational Study
Brief Title: Feeding Practices After the Surgery and Incidence of Vomiting
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Summiya Nafees Siddiqui, Professor, Aga Khan University Hospital, Pakistan
Other Study IDs: 2020-3509-11353
Record Dates: First submitted 2020-07-10; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Post-Op Complication
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is aimed to only observe the feeding practices after surgery in children undergoing below umbilicus surgery in day care and any impact of length of fasting on vomiting after surgery. If the child meets the criteria for being included in this study, the parents will be provided with informed consent form at the time of arrival at the daycare unit or at the time of arrival in the waiting area of the operating room. If parents agree and sign the consent form, then the child will be included in the study. The length of fasting period after the surgery and any episode of vomiting from after surgery till discharge time to home, will be recorded on a printed form. The nature of this study is only observation and the child will not be subjected to any new technique or medications. Parents will also be contacted on the next day of surgery on the phone number for any further observation about the child's feeding and vomiting and parental satisfaction with the anesthesia given will also be asked.

DETAILED DESCRIPTION:
After approval from the departmental research committee and College of Physicians and Surgeons Pakistan (CPSP), all pediatric patients fulfilling the inclusion criteria undergoing elective outpatient infra-umbilical surgery under general anesthesia combined with caudal analgesia at Aga Khan University Hospital would be enrolled for this study. Informed parental consent will be taken after explaining the purpose and procedure of the study.

All patients will be assessed preoperatively for anesthesia fitness by history, physical examination and laboratory investigations. On arrival on the day of surgery, patient will be premedicated with midazolam 0.3mg/kg, 30-45 minutes before the procedure. The following information including age, gender, weight, ASA status, time of last oral intake, preoperative fasting duration, surgical procedure, any history of POV with prior surgery and history of POV in parents or siblings will also be noted preoperatively. Patients at high risk of POV will not be included in the study as prophylactic antiemetic is needed to be given to such patients. Once the patient is taken into the operation room, standard ASA monitoring including electrocardiography, non-invasive blood pressure and pulse oximetry will be applied. Mode of induction will be inhalational with 8% sevoflurane and 100% oxygen or intravenous with propofol 2.5-3mg/kg. Airway will be secured with a supraglottic device appropriate to the weight of the patient. Patient will be positioned for caudal block which will be performed using small gauge butterfly cannula using 0.25% ropivacaine in a dosage of 1ml/kg body weight with a maximum safe dose of 3mg/kg. Maintenance will be achieved with isoflurane in an oxygen and nitrous oxide mixture of 60% and 40% respectively. Minimum Alveolar Concentration (MAC) will be kept between 1.0-2 %. Patients receiving any opioids or antiemetic will be excluded from the study. Intraoperative details of fluids will be noted (total volume and type of fluid). After completion of surgery, supraglottic airway device will be removed deep or awake at the discretion of primary anesthetist and patient will be shifted to the recovery. In PACU and day care ward, child will be assessed for vomiting by recording the number of episode of vomiting and for pain using Wong Baker FACES pain scale.The time of breaking NPO and type of first feed will be noted. Patient will be followed postoperatively for a period of 12 hours for any episodes of vomiting and pain in PACU and on the daycare ward. The decision of breaking NPO will be based on the current practice of pediatric surgeons and will not be interfered with.

Criteria for discharge from the PACU will include full consciousness, adequate pain control determined using Wong Baker FACES pain scale (pain score of less than 4), no bleeding, stable vital signs, and no vomiting. These patients will be followed up initially till discharge from daycare ward. Later, the child will be followed up postoperatively on second day via phone call to the parents for the occurrence of any pain and vomiting and parental satisfaction with the anesthesia will also be asked. These results will be correlated with the length of fasting.

ELIGIBILITY:
Inclusion Criteria:

* Pediatrics patients undergoing infra-umbilical elective daycare surgery under general anesthesia combined with caudal block
* Age group 2 years to 10 years
* ASA (American Society of Anesthesiologist) classification I or II

Exclusion Criteria:

* Pediatric patient who would require postoperative fasting for surgical reasons
* Patients with any known digestive pathology predisposing to post-operative vomiting (e.g. hiatal hernia and gastro-esophageal reflux)
* Patients receiving anti-emetic medications during the intraoperative period
* Patients receiving opioids during the intraoperative period

Ages: 2 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: children aged between 2-10 years of age and ASA (American Society of Anesthesiologist) classification I or II, undergoing infra-umblical daycare surgery under general anesthesia combined with caudal block will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
postoperative feeding practice | immediately after surgery to 24 hours after surgery
  adverse outcomes after restarting feeding postoperatively will be assessed

REFERENCES:
- [Background] Rizalar S, Ozbas A. Effect of Early Postoperative Feeding on the Recovery of Children Post Appendectomy. Gastroenterol Nurs. 2018 Mar/Apr;41(2):131-140. doi: 10.1097/SGA.0000000000000279. PMID 29596127
- [Background] Radke OC, Biedler A, Kolodzie K, Cakmakkaya OS, Silomon M, Apfel CC. The effect of postoperative fasting on vomiting in children and their assessment of pain. Paediatr Anaesth. 2009 May;19(5):494-9. doi: 10.1111/j.1460-9592.2009.02974.x. PMID 19453581
- [Background] Chauvin C, Schalber-Geyer AS, Lefebvre F, Bopp C, Carrenard G, Marcoux L, Mayer JF, Schwaab C, Joshi GP, Diemunsch P. Early postoperative oral fluid intake in paediatric day case surgery influences the need for opioids and postoperative vomiting: a controlled randomized trialdagger. Br J Anaesth. 2017 Mar 1;118(3):407-414. doi: 10.1093/bja/aew463. PMID 28203729
- [Background] Liechti M, Feurer R, Gross D, Schmitz A, Stutz K, Gerber A, Weiss M. Prevention of postoperative nausea and vomiting in children following adenotonsillectomy, using tropisetron with or without low-dose dexamethasone. J Anesth. 2007;21(3):311-6. doi: 10.1007/s00540-007-0523-0. Epub 2007 Aug 1. PMID 17680180
- [Background] Kranke P, Eberhart LH, Toker H, Roewer N, Wulf H, Kiefer P. A prospective evaluation of the POVOC score for the prediction of postoperative vomiting in children. Anesth Analg. 2007 Dec;105(6):1592-7, table of contents. doi: 10.1213/01.ane.0000287816.44124.03. PMID 18042855
- [Background] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for postoperative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part II. Gynecol Oncol. 2016 Feb;140(2):323-32. doi: 10.1016/j.ygyno.2015.12.019. Epub 2016 Jan 3. No abstract available. PMID 26757238
- [Background] Nelson G, Bakkum-Gamez J, Kalogera E, Glaser G, Altman A, Meyer LA, Taylor JS, Iniesta M, Lasala J, Mena G, Scott M, Gillis C, Elias K, Wijk L, Huang J, Nygren J, Ljungqvist O, Ramirez PT, Dowdy SC. Guidelines for perioperative care in gynecologic/oncology: Enhanced Recovery After Surgery (ERAS) Society recommendations-2019 update. Int J Gynecol Cancer. 2019 May;29(4):651-668. doi: 10.1136/ijgc-2019-000356. Epub 2019 Mar 15. PMID 30877144
- [Background] Shaikh SI, Nagarekha D, Hegade G, Marutheesh M. Postoperative nausea and vomiting: A simple yet complex problem. Anesth Essays Res. 2016 Sep-Dec;10(3):388-396. doi: 10.4103/0259-1162.179310. PMID 27746521
- [Background] Marulasiddappa V, Nethra HN. A Survey on Awareness about the Role of Anesthesia and Anesthesiologists among the Patients Undergoing Surgeries in a Tertiary Care Teaching Women and Children Hospital. Anesth Essays Res. 2017 Jan-Mar;11(1):144-150. doi: 10.4103/0259-1162.186595. PMID 28298774
- [Background] Thomas M, Morrison C, Newton R, Schindler E. Consensus statement on clear fluids fasting for elective pediatric general anesthesia. Paediatr Anaesth. 2018 May;28(5):411-414. doi: 10.1111/pan.13370. Epub 2018 Apr 27. PMID 29700894
- [Background] Brunet-Wood K, Simons M, Evasiuk A, Mazurak V, Dicken B, Ridley D, Larsen B. Surgical fasting guidelines in children: Are we putting them into practice? J Pediatr Surg. 2016 Aug;51(8):1298-302. doi: 10.1016/j.jpedsurg.2016.04.006. Epub 2016 Apr 21. PMID 27166876